CLINICAL TRIAL: NCT01877291
Title: Young Smokers Have Impaired Airway Defense That is Not Associated With Pulmonary Function
Brief Title: Young Smokers Have Impaired Airway Defense
Status: Completed | Type: Observational
Sponsor: University of Sao Paulo (Other)
Collaborators: Fundação de Amparo à Pesquisa do Estado de São Paulo (Other Government)
Responsible Party: Principal Investigator, Naomi Kondo Nakagawa, PT, MSc, PhD, University of Sao Paulo
Other Study IDs: CEP-FMUSP 147-13
Record Dates: First submitted 2013-06-11; First posted 2013-06-13 (Estimated); Last update posted 2013-06-17 (Estimated); Status verified 2013-06

CONDITIONS: Smoking
Keywords: smoking, nasal lavage, exhaled breath condensate, mucociliary transport
MeSH Terms: conditions — Smoking

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- Nonsmokers: Young healthy nonsmokers
- Smokers<2.5 pack years: Young "healthy" or asymptomatic smokers (aged < 35 y.o.) with smoking history <2.5 pack years
- Smokers≥ 2.5 pack-years: Young "healthy" or asymptomatic smokers (aged < 35 y.o.) with smoking history ≥ 2.5 pack-years

SUMMARY:
Background: Smoking is a key factor for development and progression of chronic obstructive pulmonary disease (COPD). Although persons with COPD often have concomitant nasal disease, there are few studies that report physiological or inflammatory changes in the upper airways in young asymptomatic smokers. The investigators investigated physiologic and inflammatory changes in the nasal and lower airways of young smokers and if these changes were related to smoking history.

Methods: Seventy-two subjects aged ≤ 35 years (32 healthy nonsmokers and 40 young smokers) participated in this study. The investigators measured nasal mucociliary clearance (MCC), nasal mucus physical properties, cell count, myeloperoxidase and cytokines concentrations in nasal lavage fluid, exhaled breath condensate (EBC) pH and lung function.

ELIGIBILITY:
Inclusion Criteria:

* healthy nonsmokers
* asymptomatic smokers
* after obtaining written informed consent

Exclusion Criteria:

* inability to understand and follow commands
* previous nasal surgery
* respiratory infection in the previous 30 days
* reported or diagnosed asthma

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Healthy nonsmokers and smokers aged between 18 and 35 y.o. that were recruited from the Faculdade de Medicina da Universidade de São Paulo
Sampling Method: Non-Probability Sample
Enrollment: 72 (Actual)
Dates: Start 2012-04; Primary Completion 2012-10 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
Exhaled Breath Condensate pH | six months

SECONDARY OUTCOMES:
mucociliary clearance by saccharine transit time test | six months

OTHER OUTCOMES:
cytokines in nasal lavage | six months

CONTACTS AND LOCATIONS:
Overall Officials: Naomi K Nakagawa, Principal Investigator — University of Sao Paulo
Locations (1):
- Faculdade de Medicina da Universidade de São Paulo, São Paulo, São Paulo, Brazil

REFERENCES:
- [Background] Rubin BK, Ramirez O, Zayas JG, Finegan B, King M. Respiratory mucus from asymptomatic smokers is better hydrated and more easily cleared by mucociliary action. Am Rev Respir Dis. 1992;145(3):545-547. Konrad F, Schreiber T, Brecht-Kraus D, Georgieff M. Mucociliary transport in ICU patients. Chest. 1994;105(1):237-241. Kim JS, Rubin BK. Nasal and sinus involvement in chronic obstructive pulmonary disease. Curr Opin Pulm Med 2008;14(2):101-104. Miller MR, Crapo R, Hankinson J, Brusasco V, Burgos F, Casaburi R, et al. General considerations for lung function testing. Eur. Respir. J. 2005;26: 153-161. Oliveira-Maul JP, de Carvalho HB, Goto DM, Maia RM, Fló C, Barnabé V, Franco DR, Benabou S, Perracini MR, Jacob-Filho W, Saldiva PHN, Lorenzi-Filho G, Rubin BK, Nakagawa NK. Aging, diabetes, and hypertension are associated with decreased nasal mucociliary clearance. Chest. 2013;143(4):1091-1097. Rubin BK, Druce H, Ramirez OE, Palmer R. Effect of clarithromycin on nasal mucus properties in healthy subjects and in patients with purulent rhinitis. Am J Respir Crit Care Med. 1997;155(6):2018-2023. Davis MD, Hunt J. Exhaled breath condensate pH assays. Immunol Allergy Clin North Am. 2012;32(3):377-386. Belda J, Parameswaran K, Keith PK, Hargreave FE. Repeatability and validity of cell and fluid-phase measurements in nasal fluid: a comparison of two methods of nasal lavage. Clin Exp Allerg. 2001;31(7):1111-1115. Koczulla AR, Noeske S, Herr C, Jörres RA, Römmelt H, Vogelmeier C, Bals R. Acute and chronic effects of smoking on inflammation markers in exhaled breath condensate in current smokers. Respiration. 2010;79(1):61-67. Nakagawa NK, Franchini ML, Driusso P, Oliveira LR, Saldiva PHN, Lorenzi-Filho G. Mucociliary clearance is impaired in acutely ill patients. Chest. 2005;128(4):2772-2777.
- [Derived] Nicola ML, Carvalho HB, Yoshida CT, Anjos FMD, Nakao M, Santos UP, Cardozo KHM, Carvalho VM, Pinto E, Farsky SHP, Saldiva PHN, Rubin BK, Nakagawa NK. Young "healthy" smokers have functional and inflammatory changes in the nasal and the lower airways. Chest. 2014 May;145(5):998-1005. doi: 10.1378/chest.13-1355. PMID 24307008